CLINICAL TRIAL: NCT02896465
Title: Treatment of Acute Childhood Diarrhoea With Human Milk Oligosaccharides and Impact on Gut Micro Biota Dysbiosis and Nutritional Status
Brief Title: Human Milk Oligosaccharides and Childhood Diarrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13.26.INF
Record Dates: First submitted 2016-08-10; First posted 2016-09-12 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Acute Diarrhea
Keywords: Children; Diarrhea; Human milk oligosaccharides
MeSH Terms: conditions — Diarrhea | interventions — World Health Organization oral rehydration solution; ORALIT; Zinc; Health Maintenance Organizations; Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ORS+ZINC (Active Comparator): Oral rehydration solution + Zinc
  Interventions: Other: Oral rehydration solution; Other: Zinc
- ORS+ZINC+HMO (Experimental): Oral rehydration solution + Zinc + Human milk oligosaccharides
  Interventions: Other: Oral rehydration solution; Other: Zinc; Other: Human milk oligosaccharides
- ORS+ZINC+Breastfeeding (Placebo Comparator): Oral rehydration solution + Zinc + Breastfeeding
  Interventions: Other: Oral rehydration solution; Other: Zinc; Other: Breastfeeding

INTERVENTIONS:
Other: Oral rehydration solution
  Other Names: ORS
Other: Zinc
Other: Human milk oligosaccharides
  Other Names: HMO
  Arms: ORS+ZINC+HMO
Other: Breastfeeding
  Arms: ORS+ZINC+Breastfeeding

SUMMARY:
Assessment of the impact of oral Human Milk Oligosaccharides (HMO) application on acute diarrhoea and the development of prolonged and persistent diarrhoea in paediatric patients hospitalized with acute diarrhoea.

DETAILED DESCRIPTION:
The trial is single site, double blind, randomized of HMO addition (1.5 g /day) to standard of care in paediatric diarrhoea patients. HMO application and follow-up of the children at home will be done for 2 weeks. Control patients receive only the standard of care (ORS plus zinc). A breastfed group of diarrhoea patients will serve as reference group.

The total sample size is 495 patients. Patients will be females and males aged 6 months to 2 years old with acute diarrhoea.

ELIGIBILITY:
Inclusion Criteria: Non breast-fed children (group I and group II):

1. Both male and female children between the ages of 6 months to 2 years.
2. Acute diarrhoea (<48 hours) without interfering co-morbidities, e.g. acute respiratory tract infection, sepsis, gross electrolyte imbalances etc.
3. Guardian is willing to have the child admitted to the hospital as an inpatient until resolution of diarrhea and to return to the clinic with the child on Day 14 after admission for a final evaluation.
4. Written informed consent must be obtained prior to admission to this study.
5. The subject has a physical examination that reveals no clinically significant abnormalities other than those expected for subjects with acute infectious diarrhea.

Exclusion Criteria: Non breast-fed children (group I and group II):

1. Children of either sex who are fully or partially breast-fed until one week before enrolment (since breastfed children receive naturally HMO, their inclusion into the ORS/zinc or HMO/ORS/zinc arms would critically interfere with the study question; depending on children's age 30 to 50 % of mothers would do so at icddr,b). However, an unblinded reference group will be constituted by age-matched children who are breastfed at the moment of hospitalization for acute diarrhea and where the mothers want to continue breastfeeding on the study ward (so breastfeeding is only an exclusion for the randomized groups).
2. Suspected or confirmed cholera as detected by a positive DF examination in stool collected on admission. (The large volume and quick evacuation of stool could interfere with product presence in the gut)
3. Symptom duration > 48 hours at screening.
4. Vomiting severity that is likely to make administration and retention of test product impossible.
5. Severe malnutrition defined (using z-scores) as: severe stunting (SS; height-for-age z-score < -3.00); severe underweight (SU; weight-for-age z-score < -3.00), and severe wasting (SW; weight-for-height z-score < -3.00), using the World Health Organization reference value. Moderate malnutrition was defined as follows: moderate stunting (height-for-age z-score -3.00 to < -2.00); moderate underweight (weight-for-age z-score -3.00 to < -2.00); and moderate wasting (weight-for-height z-score -3.00 to < -2.00). We considered children as well-nourished if their z-scores for weight-for-age, height-for-age and weight-for-height z-score were form -2.00 to +1.00.

   Children with moderate malnutrition will be enrolled since they develop with higher frequency PD).
6. Child already receiving antibiotics or anti-motility drugs for this diarrhea episode prior to screening.
7. Children with any food allergy.

Breast-fed children, (Group III - Reference group)

1. Exclusive Breastfed children Either sex: Male and female
2. Age 6-12 month
3. Acute diarrhoea (<48 hours) without interfering co-morbidities, e.g. acute respiratory tract infection, sepsis, gross electrolyte imbalances etc.
4. Written informed consent must be obtained prior to admission to this study.
5. The subject has a physical examination that reveals no clinically significant abnormalities other than those expected for subjects with acute infectious diarrhea.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 435 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Improvement (change) of clinical symptoms of diarrhea | Day1, Day2, Day3, Day4, Day5, Day6, Day7
  Passage of the last abnormal stool prior to formed/ soft stools during two consecutive 8-hour periods.

SECONDARY OUTCOMES:
Stools output | Day1, Day2, Day3, Day4, Day5, Day6, Day7
  Stools output, expressed as g/kg of body weight (cumulative output)
Weight gain | Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day14
Adverse events | Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day14
Daily stool frequency | Day1, Day2, Day3, Day4, Day5, Day6, Day7
The number of vomiting | Day1, Day2, Day3, Day4, Day5, Day6, Day7
The duration of vomiting | Day1, Day2, Day3, Day4, Day5, Day6, Day7
Change in Z-score | Day1, Day14
The amount of ORS to correct dehydration expressed as ml ORS /kg body weight, daily and cumulative input | Day1, Day2, Day3, Day4, Day5, Day6, Day7

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Diarrheal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No